CLINICAL TRIAL: NCT06631456
Title: Effects of Platelet-Rich Plasma and Ozone Therapy on Pain and Quality of Life in Knee Osteoarthritis: A Retrospective Study
Brief Title: Effects of Platelet-Rich Plasma and Ozone Therapy in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 09/07/2024-4460
Record Dates: First submitted 2024-10-05; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; platelet rich plasma; ozone therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRP group: Patients who received intra-articular PRP due to gonarthrosis
  Interventions: Other: PRP injection
- Ozone group: Patients who received intra-articular ozone therapy due to gonarthrosis
  Interventions: Other: Ozone therapy

INTERVENTIONS:
Other: PRP injection — A total of 3 doses of intra-articular PRP were applied to the symptomatic knees of the patients under ultrasound guidance, once a week.
  Groups: PRP group
Other: Ozone therapy — A total of 3 doses of intra-articular ozone therapy were applied to the symptomatic knees of the patients under ultrasound guidance, once a week.
  Groups: Ozone group

SUMMARY:
Knee osteoarthritis can frequently occur with advancing age. In cases of pain that persists despite hot/cold applications, drug therapy and exercise, intra-articular injections are considered. In advanced-stage gonarthrosis, steroid injections may respond. However, in mild and moderate knee arthritis, regenerative methods come to the forefront because the joint cartilage is still partially/completely intact. PRP and ozone therapy are frequently applied intra-articular treatments. This study will compare the effects of both injection methods on clinical outcomes.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common arthrosis that can be encountered frequently with increasing life expectancy. In mild-moderate stages, hot/cold applications, drug treatments and exercise applications are usually applied, while in those who do not respond, physical therapy or intra-articular injection treatments are applied. This retrospective study aims to examine the effects of intra-articular Platelet Rich Plasma (PRP) and ozone therapy on pain, functionality and quality of life in patients with Stage 2-3 gonarthrosis according to the Kelgren-Lawrence (KL) Classification.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years old, Stage 2-3 gonarthrosis according to KL
* Voluntariness to participate in the study

Exclusion Criteria:

* Cognitive dysfunction
* General medical condition is not suitable for injections and evaluations
* History of knee injections in the last 3 months
* History of previous knee surgery
* Bleeding disorders or those taking medications that may cause bleeding disorders after injections

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage 2-3 gonarthrosis according to KL who apply to our hospital's Physical Medicine and Rehabilitation out-patient clinic will be included.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Pain-Numerical Rating Scale | From enrollment to the end of treatment at 3rd month
  Pain level will be evaluated with the Numerical Rating Scale. (minimum: 0, maximum: 10)

SECONDARY OUTCOMES:
Pain, stiffness and physical function-WOMAC | From enrollment to the end of treatment at 3rd month
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each sub-scale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three sub-scales gives a total WOMAC score.
Quality of life-SF-12 | From enrollment to the end of treatment at 3rd month
  The 12-item short-form health survey (SF-12) quality of life scale was used to evaluate general quality of life. It was presented as a physical component score (PCS) and mental component score (MCS). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kuran, Professor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, İstanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided